CLINICAL TRIAL: NCT04076202
Title: Clinical Evaluation of Vanguard Deep Dish Rotating Platform Knee - Cementless Fixation With Finned Stem
Brief Title: Clinical Evaluation of Vanguard DD RP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU 13
Record Dates: First submitted 2019-08-23; First posted 2019-09-03 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis; Post-traumatic Osteoarthritis; Rheumatoid Arthritis
Keywords: Knee replacement; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cementless Vanguard DD RP (Experimental): Patients receiving a total knee prosthesis
  Interventions: Device: Cementless Vanguard DD RP

INTERVENTIONS:
Device: Cementless Vanguard DD RP — Patients treated with the Cementless Vanguard DD RP knee implant

SUMMARY:
This is a single cohort, prospective study of performance and safety of the Vanguard Deep Dish Rotating Platform (DD RP) cementless fixation with the goal to acquire clinical outcomes data and evaluate the performance of the device in an Austrian patient population

DETAILED DESCRIPTION:
This is a single cohort, prospective study of performance and safety of the Vanguard Deep Dish Rotating Platform (DD RP) - cementless fixation with finned stem. The performance will be assessed by Oxford Knee Score, and evaluation of aseptic loosening after 2 years follow up. Patient benefit will be evaluated by means of Knee injury and Osteoarthritis Outcome Score (KOOS) and EQ-5D patient questionnaire. The target enrollment is 113 patients in 1 clinical site in Linz, Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo primary total knee replacement:

  * with painful and disabled knee joint resulting from any of the following diagnoses:
  * Osteoarthritis,
  * Traumatic arthritis,
  * Rheumatoid arthritis with one or more compartments involved.
  * Correction of varus, valgus, or posttraumatic deformity.
  * Correction or revision of unsuccessful osteotomy or arthrodesis.
* Need to obtain pain relief and improve function.
* Ability and willingness to follow instructions, including control of weight and activity level, and to return for follow-up evaluations.
* A good nutritional state of the patient.
* Full skeletal maturity of the patient, patients who are at least 18 years of age.
* Patients of either sex.
* Consent form read, understood, and signed by patient.

Exclusion Criteria:

* Absolute contraindications include the following diagnoses:

  * Infection
  * Osteomyelitis
  * Previous partial or total prosthetic knee replacement on the operative side
  * Skeletal immaturity of the patient
  * Sepsis
  * Patients who are less than 18 years of age
* Relative contraindications include:

  * uncooperative patient or patient with neurologic disorders who are incapable of following directions,
  * osteoporosis,
  * metabolic disorders which may impair bone formation,
  * osteomalacia,
  * distant foci of infections which may spread to the implant site,
  * rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
  * vascular insufficiency, muscular atrophy, neuromuscular disease,
  * incomplete or deficient soft tissue surrounding the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2018-08-26 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance | 2 years
  The performance will be assessed by evaluation of the rate of aseptic loosening of femoral or tibial components within 2 years follow up.

SECONDARY OUTCOMES:
Patient benefits | 10 years
  Patient benefit will be evaluated by means of Knee injury and Osteoarthritis Outcome Score (KOOS). The KOOS evaluates both short-term and long-term consequences of knee injury.The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient benefits | 10 years
  Patient benefit will be evaluated by means of European Quality of Life (EuroQol) in 5 Dimensions (EQ-5D) patient questionnaire. The questionnaire contains a descriptive system and the EQ Visual Analogue scale (VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. Higher EQ-5D score values indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Illi, PhD, Study Chair — Clinical Evidence Manager; Tobias Gotterbarm, Prof. Dr., Principal Investigator — Kepler Universitäts Klinikum
Locations (1):
- Kepler Universitäts Klinikum, Linz, Austria

IPD SHARING:
Plan to Share IPD: No